CLINICAL TRIAL: NCT00492596
Title: An Evaluation of the AttenueX IntraVesical System in the Management of Female Subjects With Stress Urinary Incontinence
Brief Title: The AttenueX IntraVesical System for the Treatment of Female Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solace Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SOL2004-001
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- device (Experimental): insertion of balloon system
  Interventions: Device: AttenueX IntraVesical System
- sham (Sham Comparator): cystoscopy with sham system
  Interventions: Device: AttenueX IntraVesical System; Procedure: Sham Procedure

INTERVENTIONS:
Device: AttenueX IntraVesical System — Insertion of the Solace AttenueX Intravesical System on Day 0
  Other Names: Solace Balloon
Procedure: Sham Procedure — Cystoscopy with Simulated Insertion of AttenuEX Intravescial System
  Arms: sham

SUMMARY:
Over 11 million women in the United States suffer from stress urinary incontinence (SUI), the involuntary leakage of urine during routine physical activities such as laughing, coughing, exercising, or sneezing. SUI affects women of all ages and can result in significant emotional distress. The purpose of this study is to evaluate a non-surgical, investigational treatment intended to reduce or eliminate urine leakage due to stress urinary incontinence.

DETAILED DESCRIPTION:
A multicenter, prospective, randomized, single-blinded, two-arm longitudinal trial of the safety and effectiveness of the AttenueX Device in reducing incontinence. Subjects randomized to the control arm will have the AttenueX Device inserted at the end of the 3-month control period. For those subjects who are randomized to the treatment group, the AttenueX Device will be inserted into the bladder on Day 0, and replaced every 90 days by a new device for nine months. Subjects randomized into the treatment group will be followed for a minimum of 12 months after receiving the AttenueX Device, while subjects randomized into the control group will be followed for 3 months without the AttenueX Device and a minimum of 12 months after receiving the AttenueX Device.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 18 years of age
* Experienced stress urinary incontinence (SUI) for at least 12-months and failed prior non-surgical treatment
* VLPP ≥ 60cm H20
* Stamey Grade ≥ 1
* Free of local skin infection, impassable urethral strictures, trauma or necrosis
* Provide written informed consent

Exclusion Criteria:

* Pregnant or planning pregnancy
* 3 or more urinary tract infections within previous year
* Intrinsic sphincter deficiency
* Incontinence surgery within previous 6-months
* Cystocele ≥ grade 3
* Previous pelvic radiation therapy
* Presence of urethral abnormalities
* Recent urosepsis
* History of interstitial or follicular cystitis
* Uncontrolled diabetes
* Biofeedback within previous 3 months
* Morbid obesity
* Use of anticoagulants other than aspirin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2006-06; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Stamey Grade | 6-months

SECONDARY OUTCOMES:
Pad Weight | 6-months
VLPP | 6-months
I-QOL | 6-months
Incontinence Episode Frequency | 6-months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Arizona Urologic Specialists, Tucson, Arizona
  - Kaiser Permanente Medical Center, Downey, California
  - Tower Urology Institute for Incontinence, Los Angeles, California
  - Saad Juma Inc., San Diego, California
  - Kaiser Permanente Medical Center, San Diego, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Oak Ridge Medical Plaza, Fort Lauderdale, Florida
  - Midtown Urology, P.C., Atlanta, Georgia
  - Atlantic Health Systems, Morristown, New Jersey
  - Northeast Urogynecology, Albany, New York
  - Medical University of Southern Carolina, Charleston, South Carolina
  - Vanguard Urologic Institute, Houston, Texas
  - Integrity Medical Research, Seattle, Washington